CLINICAL TRIAL: NCT00666913
Title: Menopausal Symptoms in Women With Breast Cancer
Brief Title: Menopausal Symptoms in Women With Breast Cancer or At High Risk of Breast Cancer Treated on Another Clinical Trial
Status: Completed | Type: Observational
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CASE3107; P30CA043703 (NIH); CASE3107 (Other: Case Comprehensive Cancer Center)
Record Dates: First submitted 2008-04-24; First posted 2008-04-25 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-09

CONDITIONS: Breast Cancer; Hot Flashes
Keywords: breast cancer in situ; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; hot flashes
MeSH Terms: conditions — Breast Neoplasms; Hot Flashes; Breast Carcinoma In Situ

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: informational intervention — Data from an archived database of a closed clinical trial is retrieved.

SUMMARY:
RATIONALE: Gathering information about the frequency and intensity of hot flashes in patients with breast cancer and in patients who have a high risk of developing breast cancer may help doctors learn more about menopausal symptoms.

PURPOSE: This clinical trial is looking at menopausal symptoms in women with breast cancer or at high risk of breast cancer who received treatment on another clinical trial.

DETAILED DESCRIPTION:
OBJECTIVES:

* Retrieve data from an archived database of a closed clinical trial that involved treatment with sertraline hydrochloride or a placebo for the management of hot flashes or other menopausal symptoms in women with breast cancer or at high risk of breast cancer.
* Analyze the results of this closed clinical trial so that they can be published.

OUTLINE: Data from an archived database of a closed clinical trial is retrieved. Descriptive analyses of outcome variables (e.g., menopausal symptoms, including number and intensity of hot flashes, and psychosocial and quality of life scales) are conducted to gain insight into their distributional aspects. Data is analyzed using ANOVA with repeated measures to account for the changes within a patient over time as a function of treatment assignment. Summary scores from the psychosocial scales that are reasonably complete (i.e., FACT-B and POMS) are examined using mixed linear models to account for patient-specific differences, treatment effects, and variable patterns of completeness.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Personal or family history of carcinoma in situ of the breast or invasive breast cancer
* Treated with sertraline hydrochloride or a placebo on a clinical trial (that is now closed) at the Baylor College of Medicine-The Methodist Hospital Breast Cancer Center
* Reported hot flashes with a hot flash rating of > 15 (frequency and severity) for 1 week (before starting treatment with sertraline hydrochloride or a placebo)
* No progressive metastatic breast cancer
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Female
* Menopausal status not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data from an archived database of a closed clinical trial is retrieved.
Sampling Method: Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2007-10; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Retrieval and analysis of data regarding the frequency and intensity of hot flashes | Up to one year
  Data from an archived database of a closed clinical trial is retrieved.

SECONDARY OUTCOMES:
Assessment of psychosocial and quality of life scales (i.e., FACT-B and POMS) | Up to one year
  Summary scores from the psychosocial scales that are reasonably complete (i.e., FACT-B and POMS) are examined using mixed linear models to account for patient-specific differences, treatment effects, and variable patterns of completeness.

CONTACTS AND LOCATIONS:
Overall Officials: Lois C. Friedman, PhD, Principal Investigator — Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Locations (1):
- Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States